CLINICAL TRIAL: NCT04308915
Title: Mobile-based Games for Cognitive Training in Children With Neurodevelopmental Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indian Institute of Technology Kanpur (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IITK/IEC/2017-18II/2
Record Dates: First submitted 2020-03-11; First posted 2020-03-16 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Autism Spectrum Disorder
Keywords: digital intervention; serious games
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Game-based training (Experimental): Participants play games for cognitive training
  Interventions: Behavioral: Game-based cognitive training

INTERVENTIONS:
Behavioral: Game-based cognitive training — A suite of 5 games is presented to the participants for training working memory

SUMMARY:
Autism Spectrum Disorder (ASD) is a neurodevelopmental disorder with characteristic deficits in social functioning and presence of stereotypic behavior. Several research studies have examined potential deficits in cognitive skills, such as working memory, in this condition. A meta-analysis of the studies aimed at evaluating working memory (WM) in autistic population suggested deficits in visual and verbal aspects of WM. Working memory training has also been studied in other neurodevelopmental disorders such as Attention Deficit Hyperactivity Disorder (ADHD). The study includes development of mobile-based games for training WM and other cognitive skills in patients and the evaluation of such training in reducing symptoms of ASD. These games may also be useful for other neurodevelopmental disorders.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Autism Spectrum Disorder or another related neurodevelopmental disorder with symptoms of ASD

Exclusion Criteria:

* Inability to use smartphones/tablets
* Serious intellectual disabilities.
* Sensory impairment

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Corsi Task Block Span | change from baseline to program completion or last usage (up to 30 days of usage within 56-day trial period from the first day of data collection)
  It is an indicator of working memory. The value ranges between 0 and 9. Higher values mean better outcome.
Corsi Task Total Score | change from baseline to program completion or last usage (up to 30 days of usage within 56-day trial period from the first day of data collection)
  It is an indicator of working memory. The minimum value is 0, the maximum value has no limit. Higher values mean better outcome.

SECONDARY OUTCOMES:
Autism Treatment Evaluation Checklist Total Score | change from baseline to program completion or last usage (up to 30 days of usage within 56-day trial period from the first day of data collection)
  Autism Treatment Evaluation Checklist is a measure to evaluate treatments for Autism. The total score ranges between 0 and 179. Higher values mean better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Indian Institute of Technology Kanpur, Kanpur, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Vries M, Prins PJ, Schmand BA, Geurts HM. Working memory and cognitive flexibility-training for children with an autism spectrum disorder: a randomized controlled trial. J Child Psychol Psychiatry. 2015 May;56(5):566-76. doi: 10.1111/jcpp.12324. Epub 2014 Sep 26. PMID 25256627